CLINICAL TRIAL: NCT07095309
Title: Phase II Randomised, Double Blind, Placebo Controlled Trial of Neoadjuvant Artesunate in Stage II/III Colorectal Cancer
Brief Title: Safety and Effectiveness Study of Pre-operative Artesunate in Stage II/ III Colorectal Cancer
Acronym: NeoART-M
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Metanoic Health Ltd. (Industry)
Collaborators: Clinical Research Malaysia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-MHL-001; NMRR ID-24-01879-TSI (Other: National Medical Research Registration, Malaysia)
Record Dates: First submitted 2025-07-07; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Stage II/III Colon Cancer; Bowel Cancer
Keywords: artesunate; colorectal; drug repurposing; antimalarial
MeSH Terms: conditions — Intestinal Neoplasms | interventions — Artesunate

STUDY DESIGN:
Intervention Model Description: This is a Phase II randomised, placebo-controlled, double-blind trial of neoadjuvant oral artesunate 200 mg once daily for 14 days in patients with histologically confirmed colorectal cancer (CRC) Stage II/III awaiting surgical treatment with curative intent. The study null hypothesis is that there is no difference in survival outcomes between patients with Stage II/III colorectal cancer who receive neoadjuvant artesunate 200 mg once daily for 14 days prior to surgery and those receiving a matching placebo tablet. A randomised, placebo-controlled, double-blind design has been chosen to minimise potential researcher bias. A placebo arm is included as there is currently no standard neoadjuvant treatment in Stage II/III colon cancer.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artesuante (Experimental): Artesunate 200mg oral tablets once daily for 14 days.
  Interventions: Drug: Artesunate
- Artesunate matching placebo (Placebo Comparator): Matching placebo oral tablets once daily for 14 days.
  Interventions: Drug: Artesunate matching Placebo

INTERVENTIONS:
Drug: Artesunate — Artesunate 200mg PO OD for 14 days prior to colorectal resection surgery
  Arms: Artesuante
Drug: Artesunate matching Placebo — Matched placebo PO OD for 14 days prior to colorectal resection surgery
  Arms: Artesunate matching placebo

SUMMARY:
TThis study evaluates the safety and effectiveness of pre-operative artesunate, given orally once a day for 14 days prior to surgery, in patients with Stage II/III colorectal cancer.

Artesunate is an established antimalarial drug with an excellent safety profile. It is well tolerated, affordable, and widely available. Several laboratory studies and one small pilot clinical study in patients with colorectal cancer have shown that artesunate can reduce the proliferation and growth of cancer cells.

One hundred patients diagnosed with Stage II/III operable colorectal cancer will be randomly allocated to receive oral artesunate 200 mg daily or a matching placebo for 14 days prior to surgery. Patients will then be followed closely for 5 years to determine whether pre-operative artesunate reduces the risk of cancer recurrence after surgery.

DETAILED DESCRIPTION:
Artesunate is an established antimalarial drug belonging to the artemisinin class of drugs, has an excellent safety profile, is well tolerated and affordable. In last two decades, artemisinins have shown potent and broad anticancer properties in a range of cell lines and animal models, supporting the hypothesis that artemisinins have the potential to be an effective anti-cancer therapy. Multiple potential mechanisms of action include anti-proliferative effects through cell-cycle disruption, reactive oxygen species (ROS) -induced DNA damage, induction of apoptosis, anti-angiogenesis, immunomodulation and induced radiosensitivity.

Despite a multi-modality treatment approach to colorectal cancer, 5 year overall survival does not currently exceed 60%. Neoadjuvant pre-operative therapy may be more effective at eradicating micrometastases compared to adjuvant therapy delivered following the delay and immunological stress of surgery. However current neoadjuvant chemotherapy regimens are often associated with significant side effects and may result in a delay in surgery whilst patients recover. A well tolerated, affordable, novel anticancer agent that could be given to patients whilst they wait for surgery, without causing a surgical delay due to treatment related toxicity, would have a significant clinical impact on patient care.

The NeoART trial is a phase II multicentre randomised, double blind, placebo controlled trial (RCT) for patients undergoing primary surgery for Stage II/III colorectal cancers. Patients are randomised (1:1 ratio) to receive either a two week course of neoadjuvant artesunate 200mg once daily or matching placebo. Both patients and health care professionals are blinded to treatment allocation arm to minimise outcome-reporting bias. The primary endpoint of the trial is recurrence free survival two years after surgery. Secondary endpoints include 2 and 5 year overall survival, treatment related toxicity, tolerability and patient quality of life. A translational sub-study looking at predictive and prognostic biomarkers is also planned.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Histologically proven single primary site colorectal adenocarcinoma or high grade dysplasia plus unequivocal radiological evidence of invasive cancer
* Stage II/III colorectal cancer planned for surgical resection and no clinical indication for neoadjuvant preoperative chemotherapy/chemoradiation therapy
* WHO performance status 0,1 or 2
* Adequate full blood count: White Cell Count (WCC) >3.0 x 109 /l; Platelets >100 x 109/l; Haemoglobin (Hb) >80g/L
* Adequate renal function : Glomerular Filtration Rate >30ml/min by Cockcroft-Gault formula.
* Adequate hepatobiliary function : Total bilirubin < 3 x Upper limit norm
* Female participants of childbearing potential must have a negative pregnancy test <72 hours prior to initiating study intervention and agree to avoid pregnancy using adequate, medically approved contraceptive precautions for up to 6 weeks after the last dose of study treatment interventions.
* Male participants with a partner of childbearing potential must agree to use adequate, medically approved contraceptive precautions during and for up to 6 weeks after the last dose of the study treatment intervention.
* Patient able and willing to provide written, informed consent for the study.

Exclusion Criteria:

* Contraindication to use of artesunate due to hypersensitivity
* Pregnancy or lactation
* Male or female participants unwilling to use an effective method of birth control (either hormonal in the form of the contraceptive pill or barrier method of birth control accompanied by the use of a proprietary spermicidal foam/gel or film) ; or agreement of true abstinence from time consent is signed until 6 weeks after the last dose of study treatment intervention (i.e. withdrawal, calendar, ovulation, symptothermal and post ovulation are not acceptable methods)
* History of hearing or balance problems
* History of immunosuppression
* Patient weight < 52 kg or > 110 kg
* Other planned intervention, apart from standard of care
* Any other malignant disease diagnosis within the preceding 2 years with the exception of non-melanomatous skin cancer and carcinoma in situ
* Lactose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2032-08-30 (Estimated); Study Completion 2033-07-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) at 2 Years Post-Randomisation Assessed by Radiological and Clinical Evaluation | 2 years following study randomisation.
  RFS is defined as the time from randomisation to the first documented recurrence of colorectal cancer (local or distant) or death from any cause, whichever occurs first. Recurrence will be assessed using standard CT scans of the chest, abdomen, and pelvis, clinical examination and measuring carcinoembryonic antigen (CEA). Confirmation of recurrence may include histological evidence where clinically indicated. Unit of Measure: Months

SECONDARY OUTCOMES:
Recurrence-Free Survival at 5 Years Post-Randomisation Assessed by Radiological and Clinical Evaluation | 5 years from study randomisation
  RFS is defined as the time from randomisation to the first documented recurrence of colorectal cancer (local or distant) or death from any cause, whichever occurs first. Recurrence will be assessed using standard CT scans of the chest, abdomen, and pelvis, clinical examination and CEA . Histological confirmation of recurrence will be obtained where clinically indicated. Unit of Measure: Months
Overall Survival (OS) at 2 and 5 Years Post-Randomisation | 2 years and 5 years following study randomisation.
  Survival status will be determined through clinical follow-up, hospital records, and national death registries where available. Unit of Measure: Months
Colon Cancer-Specific Mortality at 2 and 5 Years Post-Randomisation | 2 years and 5 years following study randomisation.
Incidence of Artesunate-Related Toxicity Assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Assessment at Day 7 following initiation of study intervention (artesunate or matching placebo).
  The number of participants experiencing adverse events considered related to artesunate will be recorded and graded using the CTCAE.
  Unit of Measure:
  Number of participants with at least one artesunate-related adverse event, by CTCAE grade.
Incidence of Artesunate-Related Toxicity Assessed by Common Terminology CTCAE v5.0 | Assessment at Day 14 following initiation of study intervention (artesunate or matching placebo).
  The number of participants experiencing adverse events considered related to artesunate will be recorded and graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Causality will be assessed by the site investigator and confirmed by the clinical trial safety team. Adverse events will be coded and reported by type and severity.
Incidence of Artesunate-Related Toxicity Assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Assessment at Day 42 following initiation of study intervention (artesunate or matching placebo).
  The number of participants experiencing adverse events considered related to artesunate will be recorded and graded using the CTCAE. Causality will be assessed by the site investigator and confirmed by the clinical trial safety team. Adverse events will be coded and reported by type and severity.
  Unit of Measure:
  Number of participants with at least one artesunate-related adverse event, by CTCAE grade.
Incidence of Adverse Events Assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Assessment at Day 7 following administration of study intervention (artesunate or matching placebo).
  The number and proportion of participants experiencing any adverse events (AEs), regardless of causality, will be recorded and graded using the CTCAE.
  Unit of Measure:
  Number of participants with at least one adverse event, categorised by CTCAE grade.
Incidence Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Day 14 | Assessment at Day 14 following study intervention
  The number and proportion of participants experiencing any adverse events (AEs), regardless of causality, will be recorded and graded using the CTCAE.
  Unit of Measure:
  Number of participants with at least one adverse event, categorised by CTCAE grade.
Incidence of adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Assessment at Day 42 following study intervention
  The number and proportion of participants experiencing any adverse events (AEs), regardless of causality, will be recorded and graded using the CTCAE.
  Unit of Measure:
  Number of participants with at least one adverse event, categorised by CTCAE grade.
Pathological assessment of tumour regression post intervention | Post surgical pathology review (following Day 14 of study intervention)
  Tumour regression will be assessed by histopathological examination of the surgical resection specimen. The assessment will include:
  * Degree of tumour regression in the primary tumour bed
  * Presence of tumour involvement at the resection margins
  * Evidence of tumour invasion into the serosa (pT4a) and lymph node involvement (number and proportion of positive lymph nodes).
  * Histopathological evaluation
  Unit of Measure:
  Number and proportion of participants with positive lymph nodes, serosal involvement, and positive resection margins.
Patient-Reported Quality of Life (QoL) Assessed by Validated Questionnaires at Baseline | Assessment at Day 1 of study intervention (baseline assessment)
  Quality of life will be assessed using validated, self-administered questionnaires:
  1. EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30)
  2. EORTC QLQ-CR29 (Colorectal Cancer-Specific Module)
  These instruments evaluate global health status/QoL, functional scales (physical, role, emotional, cognitive, social), and symptom scales. Scores for each scale range from 0 to 100. For functional and global health status scales, higher scores indicate better QoL. For symptom scales, higher scores indicate worse symptoms.
  Unit of Measure:
  Mean scores for each scale/domain of the EORTC QLQ-C30 and QLQ-CR29 questionnaires.
Patient-Reported Quality of Life (QoL) Assessed by Validated Questionnaires | Assessment at Day 7 of study intervention
  Quality of life will be assessed using validated, self-administered questionnaires:
  1. EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30)
  2. EORTC QLQ-CR29 (Colorectal Cancer-Specific Module)
  These instruments evaluate global health status/QoL, functional scales (physical, role, emotional, cognitive, social), and symptom scales. Scores for each scale range from 0 to 100. For functional and global health status scales, higher scores indicate better QoL. For symptom scales, higher scores indicate worse symptoms.
  Unit of Measure:
  Mean scores for each scale/domain of the EORTC QLQ-C30 and QLQ-CR29 questionnaires.
Patient-Reported Quality of Life (QoL) Assessed by Validated Questionnaires post intervention | Assessment at Day 14 of study intervention
  Quality of life will be assessed using validated, self-administered questionnaires: 1. EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) 2. EORTC QLQ-CR29 (Colorectal Cancer-Specific Module) These instruments evaluate global health status/QoL, functional scales (physical, role, emotional, cognitive, social), and symptom scales. Scores for each scale range from 0 to 100. For functional and global health status scales, higher scores indicate better QoL. For symptom scales, higher scores indicate worse symptoms. Unit of Measure: Mean scores for each scale/domain of the EORTC QLQ-C30 and QLQ-CR29 questionnaires.
Incidence of Surgery-Related Adverse Events Assessed by CTCAE v5.0 | From time of surgery up to 3 months post surgery
  The number and proportion of participants experiencing surgery-related adverse events (AEs) will be recorded. Events will be graded using the CTCAE version 5.0, with severity classified from Grade 1 (mild) to Grade 5 (death related to AE). Events of interest include, but are not limited to, surgical site infection, anastomotic leak, wound dehiscence, postoperative bleeding, and thromboembolic events.
  Unit of Measure:
  Number of participants with at least one surgery-related AE, categorised by CTCAE grade.
Predictive value of tumour marker Carcinoma Embryonic Antigen (CEA) kinetics in terms of predicting response to artesunate therapy | Day 1 of study intervention (baseline assessment).
  Carcinoembryonic Antigen (CEA) levels will be measured in blood samples and their predictive value for response to artesunate therapy. he predictive value will be evaluated by correlating CEA with pathological tumour regression grade and recurrence-free survival.
  Unit of Measure:
  Change in serum CEA levels (ng/mL)
Predictive value of tumour marker Carcinoma Embryonic Antigen (CEA) kinetics in terms of predicting response to artesunate therapy | Assessment at Day 7 of study intervention
  Carcinoembryonic Antigen (CEA) levels will be measured in blood samples and their predictive value for response to artesunate therapy. he predictive value will be evaluated by correlating CEA with pathological tumour regression grade and recurrence-free survival.
  Unit of Measure:
  Change in serum CEA levels (ng/mL)
Predictive value of tumour marker Carcinoma Embryonic Antigen (CEA) kinetics in terms of predicting response to artesunate therapy | Assessment at Day 14 of study intervention
  Carcinoembryonic Antigen (CEA) levels will be measured in blood samples and their predictive value for response to artesunate therapy. he predictive value will be evaluated by correlating CEA with pathological tumour regression grade and recurrence-free survival.
  Unit of Measure:
  Change in serum CEA levels (ng/mL)
Predictive value of tumour marker Carcinoma Embryonic Antigen (CEA) kinetics in terms of predicting response to artesunate therapy | Assessment at Day 42 of study intervention
  Carcinoembryonic Antigen (CEA) levels will be measured in blood samples and their predictive value for response to artesunate therapy. he predictive value will be evaluated by correlating CEA with pathological tumour regression grade and recurrence-free survival.
  Unit of Measure:
  Change in serum CEA levels (ng/mL)
Immunohistochemical analyses of paraffin-embedded tumour sections to assess Kirsten rat sarcoma viral oncogene homolog (Kras) mutation status | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  KRAS mutation status will be assessed in tumour tissue sections obtained from pre-intervention (diagnostic biopsy, Day 0) and post-intervention (surgical resection, Day 15) samples. Immunohistochemistry (IHC) will be performed. Comparisons will be made to evaluate changes in mutation status and association with response to artesunate therapy.
  Unit of Measure:
  Number and proportion (%) of participants with KRAS mutant tumours at each time point.
Immunohistochemical analyses of paraffin-embedded tumour sections to assess Mismatch Repair (MMR) status | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Mismatch Repair (MMR) status will be assessed in tumour tissue sections obtained from pre-intervention (diagnostic biopsy, Day 0) and post-intervention (surgical resection, Day 15) samples. Immunohistochemistry (IHC) will be performed.
  Unit of Measure:
  Number and proportion (%) of participants with MMR-deficient tumours at each time p
Immunohistochemical analyses of paraffin-embedded tumour for v-Raf murine sarcoma viral oncogene homolog B (BRAF) mutation status | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients with BRAF mutant tumours
Immunohistochemical analyses of paraffin-embedded tumour for Platelet derived growth factor (PDGF) expression | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients whose tumours show PDGF upregulation/downregulation following treatment intervention
Immunohistochemical analyses of paraffin-embedded tumour for Vascular endothelial Growth Factor (VEGF) expression | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients whose tumours show VEGF upregulation/downregulation following study intervention
Immunohistochemical analyses of paraffin-embedded tumour on Vascular endothelial Growth Factor Receptor (VEGFR) expression | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients whose tumours show VEGFR upregulation/downregulation following study intervention
Determination of proliferative activity (Ki-67 staining, Cluster of Differentiation 31 protein (CD31) staining) | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients whose tumours show an increase or reduction in proliferation markers Ki67 and CD31 following study intervention
Determination of activation of the Deoxyribonucleic acid damage response (DDR) pathway | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients whose tumour samples show activation of the DDR pathway following study intervention
Wnt/β-catenin proliferation pathway protein expression (e.g. c-myc and cyclinD1 proteins) | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients who show an increase or a decrease in expression of proteins involved in the Wnt/β-catenin proliferation pathway (e.g. c-myc and cyclinD1 proteins) following study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Emeritus Professor Sanjeev Krishna, FRCP, ScD, FMedSci, Study Chair — Centre for Affordable Diagnotics and Therapeutics; Dr Yolanda Augustin, Principal Investigator — Centre for Affordable Diagnotics and Therapeutics
Locations (6):
- Malaysia (6):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - Pusat Perubatan Universiti Malaya, Kuala Lumpur, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Hospital Sungai Buloh, Sungai Buloh, Selangor
  - Hospital Pulau Pinang, Pulau Pinang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krishna S, Ganapathi S, Ster IC, Saeed ME, Cowan M, Finlayson C, Kovacsevics H, Jansen H, Kremsner PG, Efferth T, Kumar D. A Randomised, Double Blind, Placebo-Controlled Pilot Study of Oral Artesunate Therapy for Colorectal Cancer. EBioMedicine. 2014 Nov 15;2(1):82-90. doi: 10.1016/j.ebiom.2014.11.010. eCollection 2015 Jan. PMID 26137537
- [Background] Kremsner PG, Krishna S. Antimalarial combinations. Lancet. 2004 Jul 17-23;364(9430):285-94. doi: 10.1016/S0140-6736(04)16680-4. PMID 15262108
- [Background] Krishna S, Bustamante L, Haynes RK, Staines HM. Artemisinins: their growing importance in medicine. Trends Pharmacol Sci. 2008 Oct;29(10):520-7. doi: 10.1016/j.tips.2008.07.004. Epub 2008 Aug 25. PMID 18752857
- [Background] Schoenfeld DA. Sample-size formula for the proportional-hazards regression model. Biometrics. 1983 Jun;39(2):499-503. PMID 6354290
- [Background] Singh NP, Panwar VK. Case report of a pituitary macroadenoma treated with artemether. Integr Cancer Ther. 2006 Dec;5(4):391-4. doi: 10.1177/1534735406295311. PMID 17101767
- [Background] Steinbruck L, Pereira G, Efferth T. Effects of artesunate on cytokinesis and G(2)/M cell cycle progression of tumour cells and budding yeast. Cancer Genomics Proteomics. 2010 Nov-Dec;7(6):337-46. PMID 21156967
- [Background] Reichert S, Reinboldt V, Hehlgans S, Efferth T, Rodel C, Rodel F. A radiosensitizing effect of artesunate in glioblastoma cells is associated with a diminished expression of the inhibitor of apoptosis protein survivin. Radiother Oncol. 2012 Jun;103(3):394-401. doi: 10.1016/j.radonc.2012.03.018. Epub 2012 May 3. PMID 22560712
- [Background] Nakase I, Lai H, Singh NP, Sasaki T. Anticancer properties of artemisinin derivatives and their targeted delivery by transferrin conjugation. Int J Pharm. 2008 Apr 16;354(1-2):28-33. doi: 10.1016/j.ijpharm.2007.09.003. Epub 2007 Sep 6. PMID 17942255
- [Background] Kim SJ., Kim MS., Lee JW., Lee CH., Yoo, H., Shin, SH., et al. Dihydroartemisinin enhances radiosensitivity of human glioma cells in vitro. J Cancer Res Clin Oncol. 2006;132 :129-135. Krishna K., Ganapathi S., Ster IS., Saeed MEM., Cowan M., Finlayson C., Kovacsevics H., Jansen H., Kremsner PG., Efferth T., Kumar D. A Randomised, Double Blind,Placebo Controlled Pilot Study of Oral Artesunate Therapy for Colorectal Cancer. EBioMedicine 2015;2(1) :82-90 Kreeftmeijer-Vegter, A. R., P. J. van Genderen., Visser LG., Bierman WF., Clerinx J., van Veldhuizen CK., de Vries PJ. "Treatment outcome of intravenous artesunate in patients with severe malaria in the Netherlands and Belgium." Malar J.2012;11:102. Lai H., Nakase I., Lacoste E., Singh NP., Sasaki. Artemisinin-transferrin conjugate retards growth of breast tumors in the rat. Anticancer Res 2009;29 :3807-3810.
- [Background] Ho WE, Peh HY, Chan TK, Wong WS. Artemisinins: pharmacological actions beyond anti-malarial. Pharmacol Ther. 2014 Apr;142(1):126-39. doi: 10.1016/j.pharmthera.2013.12.001. Epub 2013 Dec 6. PMID 24316259
- [Background] Foxtrot Collaborative Group. Feasibility of preoperative chemotherapy for locally advanced, operable colon cancer: the pilot phase of a randomised controlled trial. Lancet Oncol. 2012 Nov;13(11):1152-60. doi: 10.1016/S1470-2045(12)70348-0. Epub 2012 Sep 25. PMID 23017669
- [Background] Finlay IG, Meek D, Brunton F, McArdle CS. Growth rate of hepatic metastases in colorectal carcinoma. Br J Surg. 1988 Jul;75(7):641-4. doi: 10.1002/bjs.1800750707. PMID 3416116
- [Background] Ericsson T, Blank A, von Hagens C, Ashton M, Abelo A. Population pharmacokinetics of artesunate and dihydroartemisinin during long-term oral administration of artesunate to patients with metastatic breast cancer. Eur J Clin Pharmacol. 2014 Dec;70(12):1453-63. doi: 10.1007/s00228-014-1754-2. Epub 2014 Sep 25. PMID 25248945
- [Background] Efferth T, Dunstan H, Sauerbrey A, Miyachi H, Chitambar CR. The anti-malarial artesunate is also active against cancer. Int J Oncol. 2001 Apr;18(4):767-73. doi: 10.3892/ijo.18.4.767. PMID 11251172
- [Background] Du JH, Zhang HD, Ma ZJ, Ji KM. Artesunate induces oncosis-like cell death in vitro and has antitumor activity against pancreatic cancer xenografts in vivo. Cancer Chemother Pharmacol. 2010 Apr;65(5):895-902. doi: 10.1007/s00280-009-1095-5. Epub 2009 Aug 19. PMID 19690861
- [Background] Berger TG, Dieckmann D, Efferth T, Schultz ES, Funk JO, Baur A, Schuler G. Artesunate in the treatment of metastatic uveal melanoma--first experiences. Oncol Rep. 2005 Dec;14(6):1599-603. PMID 16273263
- [Background] Berdelle N, Nikolova T, Quiros S, Efferth T, Kaina B. Artesunate induces oxidative DNA damage, sustained DNA double-strand breaks, and the ATM/ATR damage response in cancer cells. Mol Cancer Ther. 2011 Dec;10(12):2224-33. doi: 10.1158/1535-7163.MCT-11-0534. Epub 2011 Oct 13. PMID 21998290
- [Background] Beccafico S, Morozzi G, Marchetti MC, Riccardi C, Sidoni A, Donato R, Sorci G. Artesunate induces ROS- and p38 MAPK-mediated apoptosis and counteracts tumor growth in vivo in embryonal rhabdomyosarcoma cells. Carcinogenesis. 2015 Sep;36(9):1071-83. doi: 10.1093/carcin/bgv098. Epub 2015 Jul 7. PMID 26153023
- [Background] Anfosso L, Efferth T, Albini A, Pfeffer U. Microarray expression profiles of angiogenesis-related genes predict tumor cell response to artemisinins. Pharmacogenomics J. 2006 Jul-Aug;6(4):269-78. doi: 10.1038/sj.tpj.6500371. Epub 2006 Jan 24. PMID 16432535

DOCUMENTS (1):
  • Study Protocol (2024-10-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT07095309/Prot_000.pdf